CLINICAL TRIAL: NCT04870372
Title: A Multi-center, Open-Label Study to Evaluate the Efficacy and Safety of Selegiline for the Treatment of Excessive Daytime Sleepiness in Parkinson's Disease
Brief Title: Selegiline for the Treatment of Excessive Daytime Sleepiness in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2019-103-02
Record Dates: First submitted 2020-01-15; First posted 2021-05-03 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selegiline (Experimental): Subjects who meet all of the inclusion and none of the exclusion criteria will be received Selegiline.The study medication dosage will be escalated from 5mg/daily to the target dose(5~10mg/daily) in 2 weeks and then maintained for the remaining 6 weeks.
  Interventions: Drug: Selegiline

INTERVENTIONS:
Drug: Selegiline — Subjects will receive one Selegiline tablet (5 mg) per day administered at breakfast. The initial dose of Selegiline is 5 mg/day and be up-titrated in 2-week intervals in increments of 5 mg up to 10 mg (which can be taken at breakfast or divided doses of 5 mg each taken at breakfast and lunch) according to the investigator's judgment, based on individual clinical response and tolerability.
  Other Names: ELDEPRYL

SUMMARY:
This is a multi-center, open-label, single-arm 8-week investigation of Selegiline for treatment of EDS in PD patients.

DETAILED DESCRIPTION:
This is a multi-center, open-label, single-arm 8-week investigation of Selegiline. Subjects who have a diagnosis of PD based on UK brain bank criteria with ESS> 7 will be received Selegiline as an adjunctive therapy or monotherapy. This study will assess the impact of Selegiline treatment on the severity of sleep disturbances among PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and greater from 30 to 80.
2. Diagnosis of idiopathic PD according to the UK Brain Bank criteria.
3. Epworth Sleepiness Scale (ESS) >7.
4. Stable dose of anti-Parkinson drugs for at least 30 days.
5. No use of MAO-B inhibitors within the preceding 4 weeks.
6. No cognitive impairment, defined by Mini-Mental State Exam score ≤ 26.

Exclusion Criteria:

1. Diagnosis of atypical Parkinsonian syndrome, vascular Parkinsonism or drug-induced Parkinsonism.
2. Shift-work, which cannot ensure a stable sleep-wake cycle habits.
3. History of contraindications.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The mean change of ESS score will be assessed from baseline to 8 weeks when given Selegiline as an adjunctive therapy or monotherapy in PD patients with daytime sleepiness. | 8 weeks
  This outcome was used to assess relationships among changes in ESS from baseline to the endpoint.

SECONDARY OUTCOMES:
The proportion of patients with daytime sleepiness (ESS> 7) will be evaluated at the baseline and after 8 weeks treatment. | 8 weeks
  This outcome corresponds to the number of patients with daytime sleepiness.
The mean change of PDQ-8 scores will be assessed from baseline to 8 weeks of treatment. | 8 weeks
  This outcome reflects change of patients'daily quality.
The mean change of UPDRS IV items 32 and 39 scores will be assessed from baseline to 8 weeks of treatment. | 8 weeks
  This outcome corresponds to motor complications.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-feng Liu, MD,PhD, Study Chair — Second Affiliated Hospital of Soochow University
Locations (4):
- China (4):
  - Changshu Hospital Affiliated to Nanjing University of Chinese Medicine, Changshu, Jiangsu
  - Second Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiang Yuan Hospital Affiliated to Jiangsu Institute of Nuclear Medicine, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tholfsen LK, Larsen JP, Schulz J, Tysnes OB, Gjerstad MD. Development of excessive daytime sleepiness in early Parkinson disease. Neurology. 2015 Jul 14;85(2):162-8. doi: 10.1212/WNL.0000000000001737. Epub 2015 Jun 17. PMID 26085603
- [Background] Panisset M, Stril JL, Belanger M, Lehoux G, Coffin D, Chouinard S. Open-Label Study of Sleep Disturbances in Patients with Parkinson's Disease Treated with Rasagiline. Can J Neurol Sci. 2016 Nov;43(6):809-814. doi: 10.1017/cjn.2016.289. PMID 27827298